CLINICAL TRIAL: NCT03465436
Title: A Randomized, Double-blind, Placebo-controlled, 4-way Crossover Study to Compare the Effects on the Cardiac De- and Repolarization Duration as Well as Other Cardiac Safety Parameters of Two Doses of Oral Lasmiditan (100 mg and 400 mg) With Those of Moxifloxacin (400 mg) and Placebo in Healthy Subjects
Brief Title: A Study of Lasmiditan on the Heart in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16900; H8H-CD-LAHP (Other: Eli Lilly and Company); COL-MIG-105 (Other: CoLucid Pharmaceuticals); 2011-003229-88 (EudraCT Number)
Record Dates: First submitted 2018-02-05; First posted 2018-03-14 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 100 milligrams (mg) Lasmiditan (Experimental): A single, PO dose of 100 mg lasmiditan administered on Day 1 in one of four treatment periods.
  Interventions: Drug: Lasmiditan
- 400 mg Lasmiditan (Experimental): A single, PO dose of 400 mg lasmiditan administered on Day 1 in one of four treatment periods.
  Interventions: Drug: Lasmiditan
- Placebo (Placebo Comparator): Placebo for lasmiditan and placebo for moxifloxacin administered on Day 1 in one of four treatment periods.
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): A single, PO dose of moxifloxacin administered on Day 1 in one of four treatment periods.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Lasmiditan — 100 mg administered orally (PO)
  Other Names: LY573144
  Arms: 100 milligrams (mg) Lasmiditan
Drug: Lasmiditan — 400 mg administered PO
  Other Names: LY573144
  Arms: 400 mg Lasmiditan
Drug: Placebo — Placebo administered for lasmiditan or moxifloxacin
  Arms: Placebo
Drug: Moxifloxacin — 400 mg moxifloxacin administered PO
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study was to determine how two doses of lasmiditan affected the heart in healthy participants. The study also evaluated how much lasmiditan got into the blood stream and how long it took the body to get rid of it. Information about side effects was collected. The study lasted a maximum of 46 days for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within 18.5 and 29.9 kilograms per meter squared (kg/m²)
* In good physical and mental health as determined by the following:

  * Complete medical history
  * Complete physical examination
  * Vital signs including blood pressure (supine and standing), heart rate (supine and standing), respiratory rate, and temperature
  * Standard 12-lead ECG (triplicate ECG), followed by a 24-hour Holter ECG for arrhythmia monitoring
  * Clinical laboratory tests

Exclusion Criteria:

* Any of the following cardiac abnormalities on safety screening ECG:

  * QTcF interval >430 milliseconds (ms) for males, >450 ms for females
  * Unusual T wave morphology or flattened low voltage T waves
  * PR interval >240 ms or <110 ms
  * Second-degree or third-degree atrioventricular block
  * ECG evidence of complete left or right bundle branch block
  * Intraventricular conduction delay or QRS duration >110 ms
  * Supine resting heart rate <45 beats per minute (bpm) or >90 bpm
  * Pathological Q-waves
  * Evidence of ventricular pre-excitation
* Participants with a history of syncope, cardiac arrest, cardiac arrhythmia or torsade de pointes, or structural heart disease
* Participants with a family history of Long QT syndrome
* History of allergic hypersensitivity to lasmiditan or any component of the formulations
* History or current evidence of abuse of any drug substance, licit or illicit, including alcohol; a positive urine screen for drugs of abuse
* Participants with a history of postural hypotension or fainting
* Participant is not able to understand and comply with study requirements, instructions and study restrictions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2011-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants who received at least 1 dose of study drug.
Groups:
- Sequence 1 ABDC: Day 1 of each treatment period with a washout period of 7-14 days.
  A. 100 mg lasmiditan PO B. 400 mg lasmiditan PO D. 400 mg moxifloxacin PO (plus placebo) C. Placebo matched
- Sequence 2 BCAD: Day 1 of each treatment period with a washout period of 7-14 days.
  B. 400 mg lasmiditan PO C. Placebo matched A. 100 mg lasmiditan PO D. 400 mg moxifloxacin PO (plus placebo)
- Sequence 3 CDBA: Day 1 of each treatment period with a washout period of 7-14 days.
  C. Placebo matched D. 400 mg moxifloxacin PO (plus placebo) B. 400 mg lasmiditan PO A. 100 mg lasmiditan PO
- Sequence 4 DACB: Day 1 of each treatment period with a washout period of 7-14 days.
  D. 400 mg moxifloxacin PO (plus placebo) A. 100 mg lasmiditan PO C. Placebo matched B. 400 mg lasmiditan PO
Period: Period 1
Arm/Group | Sequence 1 ABDC | Sequence 2 BCAD | Sequence 3 CDBA | Sequence 4 DACB
Started | 14 | 14 | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14 | 14 | 14
Completed | 14 | 14 | 13 | 14
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1 ABDC | Sequence 2 BCAD | Sequence 3 CDBA | Sequence 4 DACB
Started | 14 | 14 | 13 | 14
Received at Least 1 Dose of Study Drug | 14 | 13 | 13 | 14
Completed | 14 | 13 | 13 | 14
Not Completed | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 ABDC | Sequence 2 BCAD | Sequence 3 CDBA | Sequence 4 DACB
Started | 14 | 13 | 13 | 14
Received at Least One Dose of Study Drug | 13 | 12 | 13 | 14
Completed | 13 | 12 | 13 | 14
Not Completed | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 ABDC | Sequence 2 BCAD | Sequence 3 CDBA | Sequence 4 DACB
Started | 13 | 12 | 13 | 14
Received at Least 1 Dose of Study Drug | 13 | 12 | 13 | 14
Completed | 13 | 12 | 12 | 14
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 ABDC | Sequence 2 BCAD | Sequence 3 CDBA | Sequence 4 DACB | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.3) | 38.4 (11.7) | 37.5 (10.8) | 40.7 (9.1) | 39.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 5 | 6 | 27
  Male | 5 | 7 | 9 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 14 | 14 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 13 | 13 | 14 | 13 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 14 | 14 | 14 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Time Matched Baseline in Mean Fridericia-Corrected QT (QTcF) Values of Lasmiditan and Moxifloxacin
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTcF = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and R-R wave (RR), which is the interval between two R waves. PR is the interval between the P wave and the ventricular depolarization wave (QRS) complex.
Time Frame: Day 1: Predose, 30 minutes postdose, 1 hour (hr), 1.5 hr, 2 hr, 2.5 hr, 3 hr, 3.5 hr, 4 hr, 6 hr, 8, hr, 12 hr and 24 hr postdose
Population: All randomized participants who received at least 1 dose of study drug and have evaluable QTcF data.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- 100 mg Lasmiditan: 100 mg lasmiditan administered PO in 1 of 4 treatment periods
- 400 mg Lasmiditan: 400 mg lasmiditan administered PO in 1 of 4 treatment periods
- Placebo: Placebo administered PO in 1 of 4 treatment periods.
- Moxifloxacin: Moxifloxacin administered PO in 1 of 4 treatment periods.
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
milliseconds
  30 minutes postdose | -8.90 (7.20) | -9.27 (6.29) | -5.49 (5.52) | 1.90 (8.69)
  1 hour postdose | -7.42 (5.83) | -4.58 (8.13) | -3.94 (5.15) | 8.36 (6.51)
  1.5 hours postdose | -7.63 (5.98) | -3.07 (7.91) | -3.68 (4.66) | 7.63 (6.32)
  2 hours postdose | -6.96 (7.08) | -1.12 (8.10) | -3.83 (5.28) | 8.16 (7.21)
  2.5 hours postdose | -5.26 (7.36) | 0.15 (8.67) | -2.89 (4.99) | 8.12 (7.15)
  3 hours postdose | -2.81 (6.95) | 2.06 (8.18) | -2.04 (5.71) | 10.01 (6.42)
  3.5 hours postdose | -2.39 (7.63) | 3.58 (6.88) | -1.85 (4.59) | 10.37 (7.09)
  4 hours postdose | -2.12 (6.89) | 4.77 (7.49) | -2.34 (5.65) | 9.39 (5.85)
  6 hours postdose | -4.33 (7.32) | -0.18 (7.38) | -3.39 (6.59) | 4.91 (7.05)
  8 hours postdose | -6.74 (7.16) | -1.84 (7.82) | -3.99 (7.11) | 3.90 (7.13)
  12 hours postdose | -3.73 (5.72) | -0.41 (6.99) | -1.79 (5.91) | 4.63 (7.12)
  24 hours postdose | 0.74 (7.51) | 0.38 (7.06) | 0.45 (6.18) | 6.61 (7.91)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -3.50, 90% CI 2-sided [-5.41 to -1.59]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -3.54, 90% CI 2-sided [-5.18 to -1.89]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -4.10, 90% CI 2-sided [-5.77 to -2.43]
Statistical Analysis 4: Comparison: 100 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -3.21, 90% CI 2-sided [-5.14 to -1.28]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.46, 90% CI 2-sided [-4.41 to -0.51]
Statistical Analysis 6: Comparison: 100 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.91, 90% CI 2-sided [-2.84 to 1.03]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.62, 90% CI 2-sided [-2.53 to 1.29]
Statistical Analysis 8: Comparison: 100 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 0.07, 90% CI 2-sided [-1.84 to 1.99]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -1.06, 90% CI 2-sided [-3.22 to 1.10]
Statistical Analysis 10: Comparison: 100 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.73, 90% CI 2-sided [-4.88 to -0.57]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.05, 90% CI 2-sided [-3.77 to -0.32]
Statistical Analysis 12: Comparison: 100 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 0.21, 90% CI 2-sided [-1.90 to 2.33]
Statistical Analysis 13: Comparison: 400 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -3.83, 90% CI 2-sided [-5.56 to -2.11]
Statistical Analysis 14: Comparison: 400 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.75, 90% CI 2-sided [-2.75 to 1.25]
Statistical Analysis 15: Comparison: 400 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 0.45, 90% CI 2-sided [-1.49 to 2.38]
Statistical Analysis 16: Comparison: 400 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 2.58, 90% CI 2-sided [0.58 to 4.58]
Statistical Analysis 17: Comparison: 400 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 2.85, 90% CI 2-sided [0.73 to 4.98]
Statistical Analysis 18: Comparison: 400 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 3.94, 90% CI 2-sided [1.85 to 6.03]
Statistical Analysis 19: Comparison: 400 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 5.28, 90% CI 2-sided [3.61 to 6.95]
Statistical Analysis 20: Comparison: 400 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 6.94, 90% CI 2-sided [4.99 to 8.89]
Statistical Analysis 21: Comparison: 400 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 3.13, 90% CI 2-sided [0.93 to 5.34]
Statistical Analysis 22: Comparison: 400 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 2.09, 90% CI 2-sided [-0.23 to 4.40]
Statistical Analysis 23: Comparison: 400 mg Lasmiditan; 12 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 1.37, 90% CI 2-sided [-0.57 to 3.30]
Statistical Analysis 24: Comparison: 400 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.29, 90% CI 2-sided [-2.21 to 1.63]
Statistical Analysis 25: Comparison: Placebo vs Moxifloxacin; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 7.32, 90% CI 2-sided [5.03 to 9.60]
Statistical Analysis 26: Comparison: Placebo vs Moxifloxacin; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 12.28, 90% CI 2-sided [10.47 to 14.10]
Statistical Analysis 27: Comparison: Placebo vs Moxifloxacin; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.27, 90% CI 2-sided [9.54 to 13.00]
Statistical Analysis 28: Comparison: Placebo vs Moxifloxacin; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.92, 90% CI 2-sided [9.97 to 13.87]
Statistical Analysis 29: Comparison: Placebo vs Moxifloxacin; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 10.98, 90% CI 2-sided [9.17 to 12.79]
Statistical Analysis 30: Comparison: Placebo vs Moxifloxacin; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.99, 90% CI 2-sided [10.10 to 13.87]
Statistical Analysis 31: Comparison: Placebo vs Moxifloxacin; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 12.19, 90% CI 2-sided [10.32 to 14.05]
Statistical Analysis 32: Comparison: Placebo vs Moxifloxacin; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.68, 90% CI 2-sided [9.83 to 13.52]
Statistical Analysis 33: Comparison: Placebo vs Moxifloxacin; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 8.24, 90% CI 2-sided [6.10 to 10.39]
Statistical Analysis 34: Comparison: Placebo vs Moxifloxacin; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 7.87, 90% CI 2-sided [5.66 to 10.07]
Statistical Analysis 35: Comparison: Placebo vs Moxifloxacin; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 6.35, 90% CI 2-sided [4.32 to 8.38]
Statistical Analysis 36: Comparison: Placebo vs Moxifloxacin; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 6.13, 90% CI 2-sided [3.88 to 8.38]

2. Secondary Outcome: Change From Time Matched Baseline in Mean Individually-Corrected QT (QTcI) Values of Lasmiditan and Moxifloxacin
Description: The corrected QT interval, individualized (QTcI) is a measurement of the electrical impulses through the largest part of the heart muscle individualized for participant pre-dose values. A negative change is a shortening of the QTc interval, a positive change is a lengthening of the QTc interval.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study drug and have evaluable QTcI data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
milliseconds
  30 minutes postdose | -9.92 (7.62) | -10.56 (8.00) | -5.27 (6.04) | 2.24 (8.88)
  1 hour postdose | -9.50 (7.74) | -6.90 (8.98) | -3.35 (5.52) | 8.96 (7.14)
  1.5 hours postdose | -9.39 (6.93) | -4.73 (8.29) | -2.81 (5.58) | 8.61 (6.42)
  2 hours postdose | -8.74 (8.34) | -2.65 (8.56) | -3.49 (5.82) | 8.29 (7.03)
  2.5 hours postdose | -7.90 (9.42) | -1.80 (8.84) | -2.44 (5.61) | 8.40 (7.53)
  3 hours postdose | -5.08 (8.29) | -0.13 (8.63) | -1.70 (6.10) | 11.01 (6.89)
  3.5 hours postdose | -3.86 (8.72) | 1.90 (7.48) | -1.67 (5.01) | 11.43 (7.38)
  4 hours postdose | -3.25 (8.07) | 3.27 (8.44) | -1.19 (6.37) | 10.28 (6.50)
  6 hours postdose | -4.84 (7.00) | -1.27 (6.65) | -3.13 (6.61) | 4.85 (7.37)
  8 hours postdose | -7.10 (7.76) | -3.08 (8.23) | -3.89 (6.77) | 4.04 (7.01)
  12 hours postdose | -4.08 (5.88) | -0.64 (6.86) | -1.65 (6.09) | 4.87 (7.14)
  24 hours postdose | 1.60 (6.84) | 0.45 (6.85) | 0.81 (6.22) | 6.74 (8.14)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -4.49, 90% CI 2-sided [-6.47 to -2.52]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -5.30, 90% CI 2-sided [-7.18 to -3.42]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -5.70, 90% CI 2-sided [-7.57 to -3.82]
Statistical Analysis 4: Comparison: 100 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -4.47, 90% CI 2-sided [-6.64 to -2.30]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -4.53, 90% CI 2-sided [-6.87 to -2.19]
Statistical Analysis 6: Comparison: 100 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.74, 90% CI 2-sided [-4.90 to -0.59]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -1.74, 90% CI 2-sided [-3.86 to 0.39]
Statistical Analysis 8: Comparison: 100 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -1.66, 90% CI 2-sided [-3.77 to 0.44]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -1.11, 90% CI 2-sided [-3.17 to 0.94]
Statistical Analysis 10: Comparison: 100 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.47, 90% CI 2-sided [-4.58 to -0.35]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.15, 90% CI 2-sided [-3.87 to -0.43]
Statistical Analysis 12: Comparison: 100 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 0.79, 90% CI 2-sided [-1.14 to 2.72]
Statistical Analysis 13: Comparison: 400 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -4.64, 90% CI 2-sided [-6.57 to -2.71]
Statistical Analysis 14: Comparison: 400 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -2.49, 90% CI 2-sided [-4.59 to -0.39]
Statistical Analysis 15: Comparison: 400 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.96, 90% CI 2-sided [-3.02 to 1.09]
Statistical Analysis 16: Comparison: 400 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 1.64, 90% CI 2-sided [-0.46 to 3.73]
Statistical Analysis 17: Comparison: 400 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 1.61, 90% CI 2-sided [-0.59 to 3.81]
Statistical Analysis 18: Comparison: 400 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 2.41, 90% CI 2-sided [0.25 to 4.57]
Statistical Analysis 19: Comparison: 400 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 4.30, 90% CI 2-sided [2.48 to 6.12]
Statistical Analysis 20: Comparison: 400 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 5.15, 90% CI 2-sided [3.02 to 7.27]
Statistical Analysis 21: Comparison: 400 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 2.77, 90% CI 2-sided [0.75 to 4.79]
Statistical Analysis 22: Comparison: 400 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 1.75, 90% CI 2-sided [-0.55 to 4.05]
Statistical Analysis 23: Comparison: 400 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = 1.75, 90% CI 2-sided [-0.19 to 3.69]
Statistical Analysis 24: Comparison: 400 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 10 milliseconds; Mixed Models Analysis; LS Mean = -0.48, 90% CI 2-sided [-2.44 to 1.48]
Statistical Analysis 25: Comparison: Placebo vs Moxifloxacin; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 7.07, 90% CI 2-sided [4.72 to 9.41]
Statistical Analysis 26: Comparison: Placebo vs Moxifloxacin; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.81, 90% CI 2-sided [9.94 to 13.69]
Statistical Analysis 27: Comparison: Placebo vs Moxifloxacin; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 10.95, 90% CI 2-sided [9.16 to 12.74]
Statistical Analysis 28: Comparison: Placebo vs Moxifloxacin; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.50, 90% CI 2-sided [9.5 to 13.43]
Statistical Analysis 29: Comparison: Placebo vs Moxifloxacin; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 10.81, 90% CI 2-sided [8.9 to 12.71]
Statistical Analysis 30: Comparison: Placebo vs Moxifloxacin; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 12.35, 90% CI 2-sided [10.42 to 14.28]
Statistical Analysis 31: Comparison: Placebo vs Moxifloxacin; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 12.65, 90% CI 2-sided [10.76 to 14.54]
Statistical Analysis 32: Comparison: Placebo vs Moxifloxacin; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 11.17, 90% CI 2-sided [9.23 to 13.10]
Statistical Analysis 33: Comparison: Placebo vs Moxifloxacin; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 8.12, 90% CI 2-sided [6.02 to 10.22]
Statistical Analysis 34: Comparison: Placebo vs Moxifloxacin; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 8.10, 90% CI 2-sided [6.01 to 10.19]
Statistical Analysis 35: Comparison: Placebo vs Moxifloxacin; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 6.26, 90% CI 2-sided [4.23 to 8.28]
Statistical Analysis 36: Comparison: Placebo vs Moxifloxacin; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 5.74, 90% CI 2-sided [3.47 to 8.01]

3. Secondary Outcome: Change From Baseline in Mean Cardiac Intervals: RR Interval of Lasmiditan and Moxifloxacin
Description: ECGs were used to calculate cardiac intervals. The RR interval is the time between two R waves.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study drug and have evaluable RR interval data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
milliseconds
  30 minutes postdose | 74.40 (76.26) | 98.52 (72.99) | 42.13 (56.00) | 18.66 (61.84)
  1 hour postdose | 149.22 (77.73) | 153.15 (65.13) | 49.87 (62.40) | 9.63 (63.32)
  1.5 hours postdose | 143.29 (80.63) | 130.79 (55.91) | 36.84 (66.52) | 13.44 (61.66)
  2 hours postdose | 118.39 (60.84) | 128.10 (48.50) | 44.69 (53.70) | 26.01 (54.44)
  2.5 hours postdose | 117.90 (73.85) | 132.86 (54.35) | 29.28 (51.39) | 26.90 (68.18)
  3 hours postdose | 105.56 (63.82) | 119.52 (60.66) | 30.84 (57.28) | 24.87 (66.41)
  3.5 hours postdose | 89.85 (56.54) | 101.86 (59.04) | 36.77 (50.34) | 19.01 (65.56)
  4 hours postdose | 72.22 (57.19) | 83.00 (56.84) | 30.32 (51.11) | 13.64 (68.55)
  6 hours postdose | -26.01 (69.03) | -3.07 (63.34) | -88.95 (60.15) | -84.12 (63.34)
  8 hours postdose | 5.63 (73.58) | 29.01 (66.89) | -50.89 (75.72) | -49.70 (52.21)
  12 hours postdose | -26.70 (77.94) | 5.19 (73.16) | -61.53 (76.51) | -74.80 (70.71)
  24 hours postdose | -16.37 (68.00) | -5.64 (63.34) | -11.66 (60.48) | -13.02 (52.97)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 32.89, 90% CI 2-sided [11.50 to 54.28]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 100.15, 90% CI 2-sided [77.81 to 122.50]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 107.11, 90% CI 2-sided [83.31 to 130.91]
Statistical Analysis 4: Comparison: 100 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 74.48, 90% CI 2-sided [56.32 to 92.63]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 89.19, 90% CI 2-sided [68.77 to 109.61]
Statistical Analysis 6: Comparison: 100 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 74.98, 90% CI 2-sided [55.41 to 94.55]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 52.83, 90% CI 2-sided [36.03 to 69.63]
Statistical Analysis 8: Comparison: 100 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 42.10, 90% CI 2-sided [24.86 to 59.35]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 62.61, 90% CI 2-sided [42.39 to 82.83]
Statistical Analysis 10: Comparison: 100 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 56.05, 90% CI 2-sided [32.49 to 79.61]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 35.71, 90% CI 2-sided [11.79 to 59.63]
Statistical Analysis 12: Comparison: 100 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.59, 90% CI 2-sided [-24.66 to 15.47]
Statistical Analysis 13: Comparison: 400 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 56.53, 90% CI 2-sided [36.72 to 76.35]
Statistical Analysis 14: Comparison: 400 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 103.30, 90% CI 2-sided [83.88 to 122.72]
Statistical Analysis 15: Comparison: 400 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 94.21, 90% CI 2-sided [75.15 to 113.26]
Statistical Analysis 16: Comparison: 400 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 83.49, 90% CI 2-sided [67.98 to 99.00]
Statistical Analysis 17: Comparison: 400 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 103.64, 90% CI 2-sided [87.28 to 120.00]
Statistical Analysis 18: Comparison: 400 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 89.26, 90% CI 2-sided [71.24 to 107.29]
Statistical Analysis 19: Comparison: 400 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 65.29, 90% CI 2-sided [48.28 to 82.30]
Statistical Analysis 20: Comparison: 400 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 52.85, 90% CI 2-sided [36.10 to 69.60]
Statistical Analysis 21: Comparison: 400 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 86.09, 90% CI 2-sided [66.36 to 105.82]
Statistical Analysis 22: Comparison: 400 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 80.12, 90% CI 2-sided [58.32 to 101.91]
Statistical Analysis 23: Comparison: 400 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 67.58, 90% CI 2-sided [44.64 to 90.51]
Statistical Analysis 24: Comparison: 400 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 7.77, 90% CI 2-sided [-10.01 to 25.55]
Statistical Analysis 25: Comparison: Placebo vs Moxifloxacin; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -22.02, 90% CI 2-sided [-38.44 to -5.60]
Statistical Analysis 26: Comparison: Placebo vs Moxifloxacin; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -38.87, 90% CI 2-sided [-57.15 to -20.60]
Statistical Analysis 27: Comparison: Placebo vs Moxifloxacin; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -22.13, 90% CI 2-sided [-39.35 to -4.91]
Statistical Analysis 28: Comparison: Placebo vs Moxifloxacin; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -17.35, 90% CI 2-sided [-32.15 to -2.56]
Statistical Analysis 29: Comparison: Placebo vs Moxifloxacin; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -1.03, 90% CI 2-sided [-18.17 to 16.12]
Statistical Analysis 30: Comparison: Placebo vs Moxifloxacin; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.77, 90% CI 2-sided [-21.81 to 12.27]
Statistical Analysis 31: Comparison: Placebo vs Moxifloxacin; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -16.56, 90% CI 2-sided [-33.36 to 0.24]
Statistical Analysis 32: Comparison: Placebo vs Moxifloxacin; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -15.29, 90% CI 2-sided [-32.94 to 2.37]
Statistical Analysis 33: Comparison: Placebo vs Moxifloxacin; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 6.13, 90% CI 2-sided [-10.86 to 23.11]
Statistical Analysis 34: Comparison: Placebo vs Moxifloxacin; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 2.27, 90% CI 2-sided [-15.25 to 19.80]
Statistical Analysis 35: Comparison: Placebo vs Moxifloxacin; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -11.95, 90% CI 2-sided [-33.46 to 9.56]
Statistical Analysis 36: Comparison: Placebo vs Moxifloxacin; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.31, 90% CI 2-sided [-17.32 to 16.69]

4. Secondary Outcome: Change From Baseline in Mean Cardiac Intervals:QRS of Lasmiditan and Moxifloxacin
Description: ECGs were used to calculate cardiac intervals. The QRS interval is the time the segment of the ECG that corresponds to depolarization of the ventricles.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study drug and have evaluable QRS data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
milliseconds
  30 minutes postdose | 0.11 (1.12) | -0.10 (1.23) | 0.09 (1.28) | -0.00 (0.97)
  1 hours postdose | -0.24 (1.21) | 0.45 (1.35) | -0.02 (1.20) | -0.12 (1.07)
  1.5 hours postdose | -0.48 (1.13) | 0.19 (1.24) | -0.37 (1.06) | -0.12 (1.09)
  2 hours postdose | -0.73 (1.12) | 0.10 (1.08) | -0.30 (1.22) | -0.29 (1.14)
  2.5 hours postdose | -0.75 (1.41) | 0.30 (1.22) | -0.21 (1.08) | -0.20 (1.11)
  3 hours postdose | -0.63 (1.21) | 0.08 (1.19) | -0.26 (1.19) | -0.35 (0.93)
  3.5 hours postdose | -0.58 (1.00) | 0.15 (1.15) | -0.17 (0.98) | -0.57 (1.34)
  4 hours postdose | -0.54 (1.03) | 0.29 (1.17) | -0.20 (0.95) | -0.58 (1.25)
  6 hours postdose | 0.20 (1.43) | 0.64 (1.50) | 0.73 (1.34) | 0.13 (1.39)
  8 hours postdose | -0.41 (1.36) | -0.39 (1.43) | -0.28 (1.38) | -0.67 (1.34)
  12 hours postdose | 0.34 (1.46) | 0.24 (1.67) | 0.63 (1.05) | 0.32 (1.52)
  24 hours postdose | 0.33 (1.22) | -0.07 (1.22) | -0.10 (1.32) | 0.09 (1.28)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.02, 90% CI 2-sided [-0.37 to 0.41]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.23, 90% CI 2-sided [-0.61 to 0.15]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.12, 90% CI 2-sided [-0.47 to 0.23]
Statistical Analysis 4: Comparison: 100 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.44, 90% CI 2-sided [-0.81 to -0.07]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.55, 90% CI 2-sided [-0.95 to -0.15]
Statistical Analysis 6: Comparison: 100 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.38, 90% CI 2-sided [-0.77 to 0.00]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.41, 90% CI 2-sided [-0.72 to -0.10]
Statistical Analysis 8: Comparison: 100 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.35, 90% CI 2-sided [-0.66 to -0.04]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.54, 90% CI 2-sided [-0.98 to -0.09]
Statistical Analysis 10: Comparison: 100 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.14, 90% CI 2-sided [-0.58 to 0.31]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.29, 90% CI 2-sided [-0.70 to 0.12]
Statistical Analysis 12: Comparison: 100 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.43, 90% CI 2-sided [0.01 to 0.84]
Statistical Analysis 13: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.19, 90% CI 2-sided [-0.59 to 0.21]
Statistical Analysis 14: Comparison: 400 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.48, 90% CI 2-sided [0.06 to 0.89]
Statistical Analysis 15: Comparison: 400 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.56, 90% CI 2-sided [0.19 to 0.93]
Statistical Analysis 16: Comparison: 400 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.40, 90% CI 2-sided [0.02 to 0.77]
Statistical Analysis 17: Comparison: 400 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.51, 90% CI 2-sided [0.13 to 0.88]
Statistical Analysis 18: Comparison: 400 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.33, 90% CI 2-sided [-0.05 to 0.71]
Statistical Analysis 19: Comparison: 400 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.32, 90% CI 2-sided [-0.02 to 0.67]
Statistical Analysis 20: Comparison: 400 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.50, 90% CI 2-sided [0.16 to 0.84]
Statistical Analysis 21: Comparison: 400 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.10, 90% CI 2-sided [-0.56 to 0.36]
Statistical Analysis 22: Comparison: 400 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.11, 90% CI 2-sided [-0.56 to 0.33]
Statistical Analysis 23: Comparison: 400 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.39, 90% CI 2-sided [-0.84 to 0.06]
Statistical Analysis 24: Comparison: 400 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.04, 90% CI 2-sided [-0.37 to 0.45]
Statistical Analysis 25: Comparison: Placebo vs Moxifloxacin; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.09, 90% CI 2-sided [-0.45 to 0.28]
Statistical Analysis 26: Comparison: Placebo vs Moxifloxacin; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.10, 90% CI 2-sided [-0.46 to 0.27]
Statistical Analysis 27: Comparison: Placebo vs Moxifloxacin; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.25, 90% CI 2-sided [-0.10 to 0.60]
Statistical Analysis 28: Comparison: Placebo vs Moxifloxacin; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.01, 90% CI 2-sided [-0.38 to 0.40]
Statistical Analysis 29: Comparison: Placebo vs Moxifloxacin; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.02, 90% CI 2-sided [-0.34 to 0.37]
Statistical Analysis 30: Comparison: Placebo vs Moxifloxacin; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.09, 90% CI 2-sided [-0.44 to 0.25]
Statistical Analysis 31: Comparison: Placebo vs Moxifloxacin; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.39, 90% CI 2-sided [-0.76 to -0.03]
Statistical Analysis 32: Comparison: Placebo vs Moxifloxacin; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.38, 90% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 33: Comparison: Placebo vs Moxifloxacin; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.60, 90% CI 2-sided [-1.03 to -0.17]
Statistical Analysis 34: Comparison: Placebo vs Moxifloxacin; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.39, 90% CI 2-sided [-0.82 to 0.04]
Statistical Analysis 35: Comparison: Placebo vs Moxifloxacin; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.31, 90% CI 2-sided [-0.70 to 0.09]
Statistical Analysis 36: Comparison: Placebo vs Moxifloxacin; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.19, 90% CI 2-sided [-0.23 to 0.61]

5. Secondary Outcome: Change From Baseline in Mean Heart Rate (HR) of Lasmiditan and Moxifloxacin
Description: Heart rate was determined during ambulatory blood pressure monitoring (ABPM).
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study drug and have evaluable HR data.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
beats per minute
  30 minutes postdose | -3.90 (5.05) | -5.51 (3.74) | -2.41 (3.22) | -1.02 (3.75)
  1 hour postdose | -7.82 (3.95) | -8.40 (3.21) | -2.77 (3.55) | -0.42 (4.05)
  1.5 hours postdose | -7.55 (4.16) | -7.41 (3.14) | -2.01 (3.53) | -0.67 (3.73)
  2 hours postdose | -6.62 (3.22) | -7.30 (2.93) | -2.65 (3.17) | -1.52 (3.19)
  2.5 hours postdose | -6.49 (4.07) | -7.59 (3.27) | -1.75 (2.97) | -1.48 (4.07)
  3 hours postdose | -5.96 (3.32) | -6.82 (3.53) | -1.83 (3.35) | -1.26 (3.95)
  3.5 hours postdose | -5.26 (3.02) | -6.02 (3.50) | -2.32 (3.06) | -0.91 (4.23)
  4 hours postdose | -4.22 (3.06) | -5.02 (3.42) | -1.82 (3.19) | -0.55 (4.37)
  6 hours postdose | 1.65 (4.52) | -0.10 (3.77) | 6.29 (5.18) | 5.84 (4.84)
  8 hours postdose | -0.43 (4.73) | -1.96 (3.93) | 3.42 (5.05) | 3.10 (3.42)
  12 hours postdose | 1.58 (5.31) | -0.50 (4.66) | 4.17 (5.46) | 4.95 (5.12)
  24 hours postdose | 1.01 (4.45) | 0.42 (4.09) | 0.89 (3.96) | 0.81 (3.60)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -1.53, 90% CI 2-sided [-2.90 to -0.16]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.09, 90% CI 2-sided [-6.29 to -3.88]
Statistical Analysis 3: Comparison: 100 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.57, 90% CI 2-sided [-6.81 to -4.32]
Statistical Analysis 4: Comparison: 100 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.01, 90% CI 2-sided [-5.00 to -3.01]
Statistical Analysis 5: Comparison: 100 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.78, 90% CI 2-sided [-5.91 to -3.65]
Statistical Analysis 6: Comparison: 100 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.14, 90% CI 2-sided [-5.20 to -3.08]
Statistical Analysis 7: Comparison: 100 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -2.94, 90% CI 2-sided [-3.87 to -2.01]
Statistical Analysis 8: Comparison: 100 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -2.42, 90% CI 2-sided [-3.42 to -1.42]
Statistical Analysis 9: Comparison: 100 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.61, 90% CI 2-sided [-6.17 to -3.06]
Statistical Analysis 10: Comparison: 100 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -3.82, 90% CI 2-sided [-5.38 to -2.26]
Statistical Analysis 11: Comparison: 100 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -2.65, 90% CI 2-sided [-4.33 to -0.97]
Statistical Analysis 12: Comparison: 100 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.12, 90% CI 2-sided [-1.22 to 1.46]
Statistical Analysis 13: Comparison: 400 mg Lasmiditan vs Placebo; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -3.09, 90% CI 2-sided [-4.16 to -2.02]
Statistical Analysis 14: Comparison: 400 mg Lasmiditan vs Placebo; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.61, 90% CI 2-sided [-6.65 to -4.58]
Statistical Analysis 15: Comparison: 400 mg Lasmiditan vs Placebo; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.39, 90% CI 2-sided [-6.42 to -4.35]
Statistical Analysis 16: Comparison: 400 mg Lasmiditan vs Placebo; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.64, 90% CI 2-sided [-5.55 to -3.72]
Statistical Analysis 17: Comparison: 400 mg Lasmiditan vs Placebo; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.82, 90% CI 2-sided [-6.77 to -4.87]
Statistical Analysis 18: Comparison: 400 mg Lasmiditan vs Placebo; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.99, 90% CI 2-sided [-6.03 to -3.96]
Statistical Analysis 19: Comparison: 400 mg Lasmiditan vs Placebo; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -3.69, 90% CI 2-sided [-4.68 to -2.71]
Statistical Analysis 20: Comparison: 400 mg Lasmiditan vs Placebo; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -3.19, 90% CI 2-sided [-4.21 to -2.17]
Statistical Analysis 21: Comparison: 400 mg Lasmiditan vs Placebo; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -6.29, 90% CI 2-sided [-7.83 to -4.95]
Statistical Analysis 22: Comparison: 400 mg Lasmiditan vs Placebo; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -5.37, 90% CI 2-sided [-6.73 to -4.02]
Statistical Analysis 23: Comparison: 400 mg Lasmiditan vs Placebo; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -4.71, 90% CI 2-sided [-6.25 to -3.17]
Statistical Analysis 24: Comparison: 400 mg Lasmiditan vs Placebo; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.55, 90% CI 2-sided [-1.74 to 0.63]
Statistical Analysis 25: Comparison: Placebo vs Moxifloxacin; 30 minutes postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 1.32, 90% CI 2-sided [0.32 to 2.33]
Statistical Analysis 26: Comparison: Placebo vs Moxifloxacin; 1 hour postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 2.29, 90% CI 2-sided [1.19 to 3.40]
Statistical Analysis 27: Comparison: Placebo vs Moxifloxacin; 1.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 1.30, 90% CI 2-sided [0.31 to 2.28]
Statistical Analysis 28: Comparison: Placebo vs Moxifloxacin; 2 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 1.07, 90% CI 2-sided [0.17 to 1.97]
Statistical Analysis 29: Comparison: Placebo vs Moxifloxacin; 2.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.21, 90% CI 2-sided [-0.81 to 1.23]
Statistical Analysis 30: Comparison: Placebo vs Moxifloxacin; 3 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.53, 90% CI 2-sided [-0.50 to 1.56]
Statistical Analysis 31: Comparison: Placebo vs Moxifloxacin; 3.5 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 1.36, 90% CI 2-sided [0.29 to 2.44]
Statistical Analysis 32: Comparison: Placebo vs Moxifloxacin; 4 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 1.21, 90% CI 2-sided [0.09 to 2.34]
Statistical Analysis 33: Comparison: Placebo vs Moxifloxacin; 6 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.49, 90% CI 2-sided [-1.97 to 0.99]
Statistical Analysis 34: Comparison: Placebo vs Moxifloxacin; 8 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.36, 90% CI 2-sided [-1.54 to 0.83]
Statistical Analysis 35: Comparison: Placebo vs Moxifloxacin; 12 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = 0.73, 90% CI 2-sided [-0.87 to 2.34]
Statistical Analysis 36: Comparison: Placebo vs Moxifloxacin; 24 hours postdose; Test type: Superiority; Mixed Models Analysis; LS Mean = -0.12, 90% CI 2-sided [-1.29 to 1.04]

6. Secondary Outcome: Number of Incidents in Electrocardiogram (ECG) Abnormalities in QTcF Interval Greater Than 450 Milliseconds
Description: ECGs were assessed for morphology abnormalities or changes in QTcf interval greater than 450 milliseconds by a board-certified cardiologist
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Incidents
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
Number analyzed (Participants) | 52 | 55 | 54 | 52
Incidents
  Predose | 0 | 0 | 0 | 0
  30 minutes postdose | 0 | 0 | 0 | 1
  1 hour postdose | 2 | 0 | 0 | 2
  1.5 hours postdose | 0 | 1 | 0 | 2
  2 hours postdose | 1 | 1 | 0 | 3
  2.5 hours postdose | 1 | 1 | 0 | 2
  3 hours postdose | 1 | 1 | 0 | 2
  3.5 hours postdose | 1 | 2 | 0 | 3
  4 hours postdose | 1 | 1 | 0 | 3
  6 hours postdose | 0 | 0 | 0 | 0
  8 hours postdose | 0 | 1 | 0 | 0
  12 hours postdose | 0 | 0 | 0 | 0
  24 hours postdose | 0 | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lasmiditan
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lasmiditan.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of lasmiditan.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan
Number analyzed (Participants) | 52 | 55
nanogram per milliliter | 104.55 (41.452) | 526.15 (240.997)

8. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC-t) of Lasmiditan
Description: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC-t) of Lasmiditan.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of lasmiditan.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan
Number analyzed (Participants) | 52 | 55
hours*nanogram per milliliter | 684.66 (278.258) | 3189.08 (1152.338)

ADVERSE EVENTS:
Time Frame: 75 days
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | 100 mg Lasmiditan | 400 mg Lasmiditan | Placebo | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55 | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/55 | 0/54 | 1/52
Other Adverse Events (participants affected / at risk) | 21/52 | 33/55 | 7/54 | 9/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Lasmiditan (N=52) | 400 mg Lasmiditan (N=55) | Placebo (N=54) | Moxifloxacin (N=52)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Lasmiditan (N=52) | 400 mg Lasmiditan (N=55) | Placebo (N=54) | Moxifloxacin (N=52)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 14 (18) | 23 (26) | 3 (4) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 5 (5) | 8 (8) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 13 (13) | 22 (22) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days